CLINICAL TRIAL: NCT01351480
Title: Assessment of Structural Benefits of Injectable Abatacept as Measured by MRI in RA Patients Who Have Failed Prior Anti-Tumor Necrosis (TNF) Therapy and Correlated With Clinical Outcomes
Brief Title: Benefits of Injectable Abatacept Using Magnetic Resonance Imaging (MRI) in Rheumatoid Arthritis (RA) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arthritis & Rheumatic Disease Specialties Research (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Norman B. Gaylis, MD, MD, Arthritis & Rheumatic Disease Specialties Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM101-306
Record Dates: First submitted 2011-05-06; First posted 2011-05-11 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Auto-immune Disease; Arthritis; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- abatacept (Other): open label use of abatacept for 12 months
  Interventions: Biological: abatacept

INTERVENTIONS:
Biological: abatacept — Abatacept administered SC weekly at 125 mg dose
  Other Names: orencia

SUMMARY:
The purpose of this study is to determine if the use of sub-cutaneous (SC) abatacept provides any structural benefit in patients with rheumatoid arthritis who have failed prior use of TNF therapy.

DETAILED DESCRIPTION:
Results in the literature suggest the structural benefits of intravenous (IV) abatacept as measured by high and low field MRI and X-ray in patients with rheumatoid arthritis who have previously failed clinical treatment with TNF agents. This study attempts to measure the structural benefits of SC abatacept in a similar cohort of patients while at the same time comparing the structural findings with clinical outcome measurements as collected at corresponding time points with an automated patient and physician disease activity scoring system of 28 joints (DAS28).

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent
* Patients must have a diagnosis of rheumatoid arthritis > 3 months
* Patients must have been receiving methotrexate for 12 weeks prior to screening at a dose of 10mg - 25 mg weekly.
* Patient must have had an inadequate response after receiving or previously receiving one (1) but no more than two (2) anti-TNF biologic agents
* Age >/= 18 yrs
* Must have active RA as defined by a DAS28 (Erythrocyte sedimentation rate) score >4.4
* Must have synovitis of at least two joints in one hand/wrist at screening and baseline
* Must have a negative Pregnancy test and use adequate method of contraception throughout the trial
* Stable use of Corticosteroids is permitted
* Stable use of Non-steroidal anti-inflammatory drugs is permitted

Exclusion Criteria:

* Functional Class IV
* Pregnancy or breastfeeding
* History of any other inflammatory arthritis
* Sexually active patients who are not using acceptable birth control
* Subjects who have undergone metacarpophalangeal (MCP) arthroplasty or anticipate the need for such a procedure
* Subjects with a history of cancer in the last five years other than non melanoma skin cancers
* Subjects who are unable to comply with study and followup procedures
* Subjects who have current or severe symptoms of renal, hepatic, hematologic, gastrointestinal, pulmonary cardiac, neurologic, or cerebral disease
* Subjects who currently abuse drugs or alcohol
* Subjects with evidence of active or latent bacterial or viral infections at the time of enrollment
* Subjects who have received live vaccines within 4 months of first dose of study medication
* Subjects with herpes zoster or cytomegalovirus that resolved less than two months prior to dosing
* Subjects at risk for tuberculosis (TB). Specifically excluded will be subjects with a history of active TB within the last 3 years and subjects with latent TB must have a negative chest X-ray and be started on treatment for at least 28 days prior to dosing.
* Prior treatment with Rituximab within 12 months
* Prior treatment with more than 2 TNFs
* Intramuscular(IM), Intravenous(IV) Intra-articular (IA) corticosteroids within 28 days prior to baseline
* Subjects who have a metal device affected by MRI (e.g. any type of electronic, mechanical or magnetic implant, metal slivers, metal objects, cardioverter defibrillator)
* Subjects who have received any disease modifying agent (DMARD) other than methotrexate within the past 28 days prior to baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman B Gaylis, MD, Principal Investigator — Arthritis & Rheumatic Disease Specialties Research
Locations (1):
- Arthritis & Rheumatic Disease Specialties Research, Aventura, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abatacept
Started | 34
Completed | 26
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Abatacept
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 6
Age, Continuous [Mean (Full Range); unit: years] | 57 [32 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Improvement in Bone Edema/Osteitis on Low-field MRI in Rheumatoid Arthritis Patients on Weekly SC Abatacept in Combination With Methotrexate Over a 12-month Period.
Description: bone edema/osteitis using low-field MRI analysis of 25 anatomical locations in the wrist and hand and scoring the volume of the original articular bone in 0.5 increments from 0-3, with each increment in the scale representing 33% of the volume of the peripheral 1 cm of original (eroded + residual) articular bone.
Time Frame: MRIs at Baseline and Week 48
Population: osteitis on the MRIs from 27 patients at baseline and week 48
Measure: Number; unit: participants
Arm/Group | Abatacept
Number analyzed (Participants) | 27
participants | 27

2. Secondary Outcome: Patients With an Improvement in DAS Score Were Considered Responders at Week 48
Description: Patient with a positive change in DAS score were considered responders . The DAS score is calculated using the number of tender and swollen joints based upon a 28 joint count, the ESR in mm/hr., and the physician global score
Time Frame: The DAS 28 score will be performed at baseline and 48
Population: There were 34 enrolled patients with 7 patients who early termed so analysis was performed on 27 patients
Measure: Number; unit: participants
Arm/Group | Abatacept
Number analyzed (Participants) | 27
participants | 25

3. Secondary Outcome: To Measure the Change From Baseline in Patient DAS 28 Scores at Baseline and Weeks 12, 24
Description: DAS 28> 5.1=high disease activity DAS28 <3.2=low disease activity DAS28 <2.6=remission Criteria used in formula are number of tender joints based upon 28 joints, number of swollen joints based on 28 joints, ESR in mm/hr and patient global health core based on 0-10 mm
Time Frame: Patient DAS 28 scores will be measured at baseline and weeks 12, 24, 48 and disease activity will be recorded at Week 48
Population: the number of participants who reached remission, low disease activity, moderate disease activity and high disease activity will be determined as based upon the DAS scale
Measure: Number; unit: participants
Arm/Group | Abatacept
Number analyzed (Participants) | 27
participants
  clinical remission at week 12 | 2
  low disease activity at week 12 | 2
  mod disease activity at week 12 | 12
  high disease activity at week 12 | 11
  clinical remission at week 24 | 1
  low disease activity at week 24 | 2
  moderate disease activity at week 24 | 14
  high disease activity at week 24 | 8
  clinical remission at week 48 | 4
  low disease activity at week 48 | 6
  moderate disease activity at week 48 | 8
  high disease activity at week 48 | 7

4. Secondary Outcome: the Clinical Outcomes Measurements (American College of Rheumatology Activity Scoring, Health Assessment The Number of Patients With a Clinical Response at Week 24 and 48
Description: Patient with a positive change in DAS score were considered responders . The DAS score is calculated using the number of tender and swollen joints based upon a 28 joint count, the ESR in mm/hr., and the physician global score (1-10 cm). Total maximum score was at high disease activity at baseline.
Time Frame: week 24 and Week 48
Population: There were 34 enrolled patients with 7 patients who early termed so analysis was performed on 27 patients
Measure: Number; unit: participants
Arm/Group | Abatacept
Number analyzed (Participants) | 27
participants
  clinical response at 6 months | 20
  clinical response at 12 months | 25

5. Secondary Outcome: Number of Patients With Adverse Events
Description: site will report the number of patients with adverse envents from Day 1 up to 52 weeks
Time Frame: all adverse events will be captured from Day 1 up to 52 weeks
Population: There were 34 enrolled patients with 7 patients who early termed so analysis was performed on 27 patients
Measure: Number; unit: participants
Arm/Group | Abatacept
Number analyzed (Participants) | 27
participants | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Abatacept
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes